CLINICAL TRIAL: NCT01749696
Title: Alterations in Connective Tissue in Patients With or Without Pelvic Organ Prolapse.
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 33/180/2009
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Connective tissue; Elastin; Collagen
MeSH Terms: conditions — Pelvic Organ Prolapse; Aortic Stenosis, Supravalvular

GROUPS / COHORTS (2):
- Patients with pelvic organ prolapse: Patients, who were operated on because of pelvic organ prolapse.
- Patients without pelvic organ prolapse: Patients, who had hysterectomy due to other reasons than pelvic organ prolapse.

SUMMARY:
The aim of our study is to investigate the alterations in connective tissue of vaginal wall in patients with and without pelvic organ prolapse (POP).

DETAILED DESCRIPTION:
The tissue samples were taken from the anterior wall of vagina in the midline close to cervix or apex. The tissue samples were collected from the vaginal wall of the patients with pelvic organ prolapse (n=39) during vaginal prolapse surgery. Control samples (n=39) were taken from patients after vaginal or laparoscopic removal of the uterus.

The formalin-fixed and paraffin embedded tissue samples were stained with Verhoeff van Gieson and Movat's pentachrome. Samples were examined by pathologist and gynecologist blinded as to the other investigator and to the pelvic organ prolapse status. In case of discrepancy investigators evaluated the samples together to gain consensus.

ELIGIBILITY:
Inclusion Criteria:

* surgery for pelvic organ prolapse
* hysterectomy due to other benign reasons than pelvic organ prolapse

Exclusion Criteria:

* surgery due to malignancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 39 patients with pelvic organ prolapse and as controls 39 patients without prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The elastin content in tissue samples in patients with or without pelvic organ prolapse. | september 2012

SECONDARY OUTCOMES:
The collagen content in tissue samples in women with or without pelvic organ prolapse. | September 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Turku University Central Hospital, Turku, Finland